CLINICAL TRIAL: NCT06610747
Title: Home Care Monitoring of Visual Acuity and OCT Versus Standard Hospital/Clinic Care Monitoring During Diabetic Macular Edema Management: A Non-inferiority Randomized Clinical Trial
Brief Title: Home- vs Hospital-based Care of Anti-VEGF Treatment for Diabetic Macular Edema: Non-inferiority RCT
Acronym: DME HOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: Dongguan Guangming Ophthalmic Hospital (Unknown); The Second People's Hospital of Foshan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024KYPJ072
Record Dates: First submitted 2024-08-27; First posted 2024-09-24 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic macular edema; Diabetic retinopathy; Aflibercept; Anti-VEGF; Home care monitoring; Home OCT; Best-corrected visual acuity; Visit burden; Randomized clinical trial
MeSH Terms: conditions — Diabetic Retinopathy | interventions — aflibercept; Laser Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home-based care group (Experimental): Home-based monitoring with home visual acuity tester and home OCT:
  For participants in the home-based care group, home service appointments will be scheduled during the 'pro re nada' (PRN) treatment phase. Participants will receive a home self-administered visual acuity tester and a self-administered Home OCT to use at home every 4 weeks after the 5th injection through 48 weeks, and then as needed per the DME treatment regimen protocol provided in the protocol.
  Interventions: Procedure: Home-based Care Monitoring; Drug: Aflibercept 2Mg/0.05Ml Inj,Oph; Procedure: Laser Treatment
- Standard Hospital/clinic-based care group (Active Comparator): Standard hospital/clinic-based visual acuity and OCT monitoring:
  For participants in the standard Hospital/clinic-based group, hospital service appointments will be scheduled during the 'pro re nada' (PRN) treatment phase. Participants will be instructed to return to the clinic for hospital-based visual acuity examinations and standard OCT measurements every 4 weeks after the 5th injection through 48 weeks, and then as needed per the DME treatment regimen protocol provided in the protocol.
  Interventions: Drug: Aflibercept 2Mg/0.05Ml Inj,Oph; Procedure: Laser Treatment; Procedure: Standard Hospital/clinic-based Care Monitoring

INTERVENTIONS:
Procedure: Home-based Care Monitoring — For participants in the home-based care group, home service appointments will be scheduled during the 'pro re nada' (PRN) treatment phase. Participants will receive a home self-administered visual acuity tester and a self-administered Home OCT to use at home every 4 weeks after the 5th injection through 48 weeks, and then as needed per the DME treatment regimen protocol provided in the protocol. The results of the visual acuity and OCT measurements will be transmitted to the clinician at the hospital. An online discussion between the clinician and the participant will be held. Reports will be sent to the participant after each visit. In the event that the study coordinator is unable to contact the participant, a total of three phone call attempts will be made. Any failure to keep an appointment will be communicated to the participant.
  Arms: Home-based care group
Drug: Aflibercept 2Mg/0.05Ml Inj,Oph — Each eye will receive three to five q4week loading anti-VEGF injections of aflibercept (2-mg, EYLEA®) after enrollment to complete the initial loading phase of 5 doses. Each eye will then be treated according to the PRN treatment protocol described in the study protocol.
  Other Names: Aflibercept 2-mg/0.05mL intravitreal ophthalmic injection
Procedure: Laser Treatment — Panretinal photocoagulation (PRP) may be administered if deemed necessary by the investigator, typically for high-risk proliferative diabetic retinopathy (PDR). However, individuals are not eligible for this study if it is expected that they will require PRP within 6 months at the time of enrollment. In general, PRP should not be given to study participants with less than high risk PDR. For previously untreated eyes exhibiting PDR with high-risk characteristics, PRP should be administered promptly, while it can be considered, although generally not recommended, for persons with non-high-risk PDR or severe non-PDR who are being monitored monthly in this protocol. Focal/grid laser typically should be withheld until sometime after the final visit.
Procedure: Standard Hospital/clinic-based Care Monitoring — For participants in the standard Hospital/clinic-based group, hospital service appointments will be scheduled during the &#39;pro re nada&#39; (PRN) treatment phase. Participants will be instructed to return to the clinic for hospital-based visual acuity examinations and standard OCT measurements every 4 weeks after the 5th injection through 48 weeks, and then as needed per the DME treatment regimen protocol provided in the protocol. A discussion between the clinician and the participant will be held in clinic. Reports will be sent to the participant after each visit. In the event that the study coordinator is unable to contact the participant, a total of three phone call attempts will be made. Any failure to keep an appointment will be communicated to the participant.
  Arms: Standard Hospital/clinic-based care group

SUMMARY:
Diabetic macular edema (DME) is a common cause of central visual loss in diabetic patients and a global public health burden around the world. Most patients with DME and vision loss require pharmacological inhibition using anti-VEGF agents with multiple monitoring visits that require both visual acuity testing and optical coherence tomography (OCT) to determine if re-treatment is warranted as well as the recommended time interval to the next follow-up visit. However, this treatment regimen often requires monthly or every other month clinic visits, which places a substantial burden on ophthalmic clinics and patients.

Recently, portable self-administered Home OCT devices have been developed that allow for home-based OCT scanning of retinal diseases, e.g., DME, although these devices do not include visual acuity determination. The investigators previously proposed to deliver Home OCT devices and Home visual acuity tester to patients' homes to complete routine monitoring visits at home. However, there is a lack of evidence regarding the safety and efficacy of this novel monitoring regimen for DME patients, specifically whether its use could reduce the burden associated with frequent hospital visits without sacrificing visual acuity outcomes.

This study aims to provide evidence to support use of a novel monitoring regimen for DME patients that could substantially reduce the burden associated with frequent hospital visits without sacrificing visual acuity outcomes.

DETAILED DESCRIPTION:
This visit and treatment burden is associated with poorer DME treatment outcomes in the clinical practice (real world) setting compared with outcomes in clinical trials. Studies have shown that less than half of DME patients remain compliant with their anti-VEGF treatment schedules in the clinical practice setting, with many experiencing worse visual acuity levels after missed appointments. Potential reasons for suboptimal outcomes include under-treatment when otherwise indicated, missed visits when treatment should be applied, absence of protocol refractions and protocol visual acuity measurements which may guide treatment but be difficult to obtain in clinic, and anti-VEGF costs. Addressing these challenges could benefit from a novel approach of monitoring patients remotely so that visits only would be needed when treatment was warranted based on changes in best corrected visual acuity or OCT central subfield thickness measurements, but only if this approach does not sacrifice visual acuity outcomes. In particular, reducing the frequency of clinic visits might improve patient compliance and potentially improve treatment outcomes.

To address these challenges, new devices, which currently are not readily available around the world, and new agents or anti-VEGF delivery devices have been developed to try to reduce the burden of injections without sacrificing visual acuity outcomes. However, most of these new agents that could be given q8 or q12 or q16 weeks in some study participants provided non-inferior visual acuity outcomes only in the setting of protocols that included q4week clinic assessments. Potentially, this frequent monitoring may be needed to avoid sacrificing visual acuity outcomes when reducing the number of injections. Furthermore, new delivery devices have been fraught with safety concerns.

Recently, portable self-administered Home OCT devices have been developed that allow for home-based OCT scanning of retinal diseases, e.g., DME, nAMD, or CNV associated with pathologic myopia. The image quality and accuracy of retinal thickness measurements obtained from some of these devices have been validated through comparison with clinic- or hospital-based OCTs, although evaluation of these devices has not included home monitoring of visual acuity, nor determined if their use results in non-inferior visual acuity outcomes.

In this study, the investigators will conduct a non-inferiority randomized clinical trial to determine if the mean change in visual acuity (primary outcome) is non-inferior with the home monitoring of visual acuity and OCT compared with hospital/clinic-based care among DME participants receiving anti-VEGF therapy, and if it is non-inferior, to determine if the home care model can reduce hospital/clinic visits over 96 weeks (principal secondary outcome).

Participants will receive five q4week loading anti-VEGF injections after enrollment. Only those participants who receive loading injections as planned will be assigned randomly to one of two groups and undergo as needed (pro-re-nata, PRN) treatments with injections of anti-VEGF:

1. Home-based Care Group
2. Standard Hospital/clinic-based Care Group

Re-injections of anti-VEGF (PRN), laser, surgery or other procedures will be performed per protocol for participants from both groups.

ELIGIBILITY:
Participant-level Criteria:

Inclusion Criteria:

To be eligible, the following inclusion criteria must be met:

* Age of 18 years or older;
* Type 1 or type 2 diabetes mellitus
* Current regular use of insulin for the treatment of diabetes or current regular use of oral anti-hyperglycemia agents for the treatment of diabetes
* Travel time from home to the hospital/clinic within a 2-hour driving distance
* At least one eye meets the study eye criteria listed in Section 2.4
* Ability and willingness to operate the self-administrated visual acuity tester and Home OCT device by themselves or with the help of family after training
* Ability and willingness to provide informed consent

Exclusion Criteria:

An individual is not eligible if any of the following exclusion criteria are present:

* Conditions that would preclude participation in the study, such as unstable medical status including blood pressure, cardiovascular disease, renal disease, and glycemic control as determined by the investigators
* History of systemic anti-VEGF or pro-VEGF treatment within 4 months before randomization. These drugs should not be used during the study;
* In an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval for the indication being studied
* Blood pressure > 180/110 (systolic above 180 or diastolic above 110. If blood pressure is brought below 180/110 by anti-hypertensive treatment, then the individual may be eligible
* History of myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months before enrollment
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 2 years. Women who are potential study participants should be questioned about the potential for pregnancy, and the investigator will determine when a pregnancy test is needed
* Currently participating in other clinical trials
* The individual who might move out to an area beyond 2-hour driving distance during the first 12 months of the study

Study eye-level Criteria:

The participant must have at least one eye meeting all of the inclusion criteria and none of the exclusion criteria listed below. Participants can have only one study eye. If both eyes are eligible at the time of enrollment and one of the eyes has never received anti-VEGF treatment, that eye should be included. If both eyes are eligible and have previously received anti-VEGF treatment or both eyes have never received anti-VEGF, then the better-seeing eye will be selected before enrollment. If neither eligible eye is the better-seeing eye, then the investigator and participant will select the study eye by mutual agreement before enrollment.The definition of better-seeing, worse-seeing and same eye is in the followings:

* If the baseline visual acuity letter score in both eyes is 50 (20/100) or better, the better-seeing eye is the eye with better baseline visual acuity (better than that of the fellow eye by 5 letters or more), and the worse-seeing eye is the eye with worse baseline visual acuity (worse than that of the fellow eye by 5 letters or more); if the baseline visual acuity of one eye is within 4 letters of that of the fellow eye, the two eyes are the same and neither eye is the better-seeing eye.
* If the baseline visual acuity letter score in both eyes is < 50 (20/100), the better-seeing eye is the eye with better baseline visual acuity (better than that of the fellow eye by 10 letters or more), and the worse-seeing eye is the eye with worse baseline visual acuity (worse than that of the fellow eye by 10 letters or more); if the baseline visual acuity of study eye is within 9 letters of that of the fellow eye, the two eyes are the same and neither eye is the better-seeing eye.

The eligibility criteria for a study eye are as follows:

Inclusion Criteria:

* Central-involved DME (central subfield thickness on OCT defined on Heidelberg Spectralis OCT 320 μm or more in men and 305 μm or more in women, or Zeiss Cirrus OCT 305 μm or more in men and 290 μm or more in women, or the equivalent on spectral-domain OCT based on gender specific cutoffs)
* Best corrected visual acuity letter score ≤ 78 (i.e., 20/32 or worse) and ≥ 24 (i.e., 20/320 or better) within seven days of inclusion
* Received no treatment for DME before, or received no anti-VEGF injection for DME within the past 3 months; however, if there is a history of anti-VEGF injections, <=1 injection in the past year and <=3 injections over the study participant's lifetime); or, <=2 monthly injections within the past 3 months and <=3 injections over the past year, and <=6 injections over the study participant's lifetime.
* Sufficient media clarity, pupillary dilation, and individual cooperation to allow for adequate fundus photographs and adequate OCT

Exclusion Criteria:

The following exclusions apply to the study eye only (i.e., they may be present for the non-study eye):

* Macular edema due to reasons other than diabetes
* Any history of prior laser, other surgical or corticosteroid treatment for DME (such as focal/grid macular photocoagulation, intravitreal corticosteroids or peribulbar corticosteroids) within the prior 12 months
* History of intravitreal anti-VEGF for an ocular condition other than DME (e.g., choroidal neovascularization, central retinal vein occlusion, PDR) within the prior 6 months or anticipated need in the next 6 months
* Coexisting ocular diseases that might alter visual acuity during the course of the study, such as a retinal vein or artery occlusion, uveitis or other ocular inflammatory diseases, neovascular glaucoma, etc.
* A substantial cataract that, in the investigator's opinion, is likely to be decreasing visual acuity by 3 lines or more. This means that the cataract would be reducing acuity to 20/40 or worse if the eye were otherwise normal
* History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckling, any intraocular surgery, etc.) within prior 4 months or anticipated within the next 6 months following randomization
* Uncontrolled glaucoma
* Severe external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in best-corrected visual acuity (letter score) in the study eyes from the randomization visit to 96 week visit | From the randomization visit to 96 week visit
  The randomization visit is defined as the visit of the 5th loading dose. Best-corrected visual acuity (letter score) will be measured by masked optometrists using the ETDRS tumbling-E eye chart. The testing procedures are detailed in the study protocol.

SECONDARY OUTCOMES:
Hospital/clinic visits with the home-based care group versus standard hospital/clinic-based care group | from the randomization visit to 96 week visit
  Hospital/clinic visits for DME or DR is the principal secondary outcome.
Proportion of study eyes with at least 5, 10 and 15 letter gains or losses in visual acuity | from the randomization visit to 96 week visit
  Proportion of study eyes with at least 5, 10 and 15 letter gains or losses in visual acuity from the randomization visit to 96 week visit. Distribution of visual acuity outcomes (20/20 or better; 20/25 or better; 20/40 or better; 20/80 or better; 20/200 or better) will also be described.
Change in OCT central subfield thickness | from the randomization visit to 96 week visit
  OCT examinations will be conducted by masked, experienced technicians. The same machine type should be used throughout the study for each participant. The outcomes include change in OCT central subfield thickness and retinal volume.
Change in OCT retinal volume | from the randomization visit to 96 week visit
  OCT examinations will be conducted by masked, experienced technicians. The same machine type should be used throughout the study for each participant. The outcomes include change in OCT central subfield thickness and retinal volume.
Long lapses in care | from the randomization visit to 96 week visit
  Lapse in care will be defined as more than 2 weeks past the target date for a visit that is scheduled either 4 or 8 weeks after a completed visit or more than 4 weeks past the target date for a visit scheduled 16 or more weeks after a completed visit. Detailed definition is provided in the protocol.
Ability to Work and Perform Regular Activities | from the randomization visit to 96 week visit
  The Work Productivity and Activity Impairment Questionnaire Global Health (WPAI-GH, Simplified Chinese version) will be used to evaluate the ability to work and perform regular activities. The WPAI-GH is a validated survey tool that consists of 6 questions assessing the impact of health problems on work performance and on regular daily activities outside of work.

OTHER OUTCOMES:
Economic analysis (Cost-utility ratio) | from the randomization visit to 96 week visit
  Costs and Utilities will be calculated over the duration of the trial. The incremental cost-utility ratio (ICUR) will be calculated by taking the incremental cost of the home-based care model over the hospital/clinic-based care model and dividing them by the incremental utilities of home-based care model over hospital/clinic-based care model. A probabilistic sensitivity analysis will be conducted to better characterize overall uncertainty in the results. Details are provided in the statistical analysis protocol (SAP).
Change in best-corrected visual acuity (letter score) in the non-study eyes from the randomization visit to 96 week visit | From the randomization visit to 96 week visit
  The randomization visit is defined as the visit of the 5th loading dose. Best-corrected visual acuity (letter score) will be measured by masked optometrists using the ETDRS tumbling-E eye chart. The testing procedures are detailed in the study protocol. Data in the non-study eyes will be analyzed.
Change in best-corrected visual acuity (letter score) in the study eyes from the randomization visit to 48 week visit | From the randomization visit to 48 week visit
  The randomization visit is defined as the visit of the 5th loading dose. Best-corrected visual acuity (letter score) will be measured by masked optometrists using the ETDRS tumbling-E eye chart. The testing procedures are detailed in the study protocol. Proportion of study eyes with at least 5, 10 and 15 letter gains or losses in visual acuity, distribution of visual acuity outcomes (20/20 or better; 20/25 or better; 20/40 or better; 20/80 or better; 20/200 or better) from the randomization visit to 48 week visit will also be described.
Change in OCT retinal volume from the randomization visit to 48 week visit | from the randomization visit to 48 week visit
  OCT examinations will be conducted by masked, experienced technicians. The same machine type should be used throughout the study for each participant. The outcomes include change in OCT central subfield thickness and retinal volume.
Change in OCT central subfield thickness from the randomization visit to 48 week visit | from the randomization visit to 48 week visit
  OCT examinations will be conducted by masked, experienced technicians. The same machine type should be used throughout the study for each participant. The outcomes include change in OCT central subfield thickness and retinal volume.
Long lapses in care from the randomization visit to 48 week visit | from the randomization visit to 48 week visit
  Lapse in care will be defined as more than 2 weeks past the target date for a visit that is scheduled either 4 or 8 weeks after a completed visit or more than 4 weeks past the target date for a visit scheduled 16 or more weeks after a completed visit. Detailed definition is provided in the protocol.
Ability to Work and Perform Regular Activities from the randomization visit to 48 week visit | from the randomization visit to 48 week visit
  The Work Productivity and Activity Impairment Questionnaire Global Health (WPAI-GH, Simplified Chinese version) will be used to evaluate the ability to work and perform regular activities. The WPAI-GH is a validated survey tool that consists of 6 questions assessing the impact of health problems on work performance and on regular daily activities outside of work.
Change in superficial capillary vessel density (SVD) in the study eyes | Baseline, 4, 8, 12, 16 (randomization), 24, 48, 72, 96 week visit
  The vessel density of the superfcial capillary plexus level will be analyzed in the 3x3 mm OCTA scanning mode (Zeiss Cirrus HD-OCT).
Change in deep capillary vessel density (DVD) in the study eyes | Baseline, 4, 8, 12, 16 (randomization), 24, 48, 72, 96 week visit
  The vessel density of the deep capillary plexus level will be analyzed in the 3x3 mm OCTA scanning mode (Zeiss Cirrus HD-OCT).
Change in foveal avascular zone (FAZ) in the study eyes | Baseline, 4, 8, 12, 16 (randomization), 24, 48, 72, 96 week visit
  The area of foveal avascular zone will be analyzed in the 3x3 mm OCTA scanning mode (Zeiss Cirrus HD-OCT).
Change in non-perfusion (NP) in the study eyes | Baseline, 4, 8, 12, 16 (randomization), 24, 48, 72, 96 week visit
  The NP regions in the superficial and deep capillary plexus were will be evaluated on the 3x3 mm OCTA Image.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, MD, PhD, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (3):
- China (3):
  - Dongguan Guangming Ophthalmic Hospital, Dongguan, Guangdong
  - The Second Peoples Hospital of Foshan, Foshan, Guangdong
  - State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reddy RK, Pieramici DJ, Gune S, Ghanekar A, Lu N, Quezada-Ruiz C, Baumal CR. Efficacy of Ranibizumab in Eyes with Diabetic Macular Edema and Macular Nonperfusion in RIDE and RISE. Ophthalmology. 2018 Oct;125(10):1568-1574. doi: 10.1016/j.ophtha.2018.04.002. Epub 2018 May 8. PMID 29752001
- [Background] Jhaveri CD, Glassman AR, Ferris FL 3rd, Liu D, Maguire MG, Allen JB, Baker CW, Browning D, Cunningham MA, Friedman SM, Jampol LM, Marcus DM, Martin DF, Preston CM, Stockdale CR, Sun JK; DRCR Retina Network. Aflibercept Monotherapy or Bevacizumab First for Diabetic Macular Edema. N Engl J Med. 2022 Aug 25;387(8):692-703. doi: 10.1056/NEJMoa2204225. Epub 2022 Jul 14. PMID 35833805
- [Background] Heier JS, Korobelnik JF, Brown DM, Schmidt-Erfurth U, Do DV, Midena E, Boyer DS, Terasaki H, Kaiser PK, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Vitti R, Berliner AJ, Zeitz O, Metzig C, Holz FG. Intravitreal Aflibercept for Diabetic Macular Edema: 148-Week Results from the VISTA and VIVID Studies. Ophthalmology. 2016 Nov;123(11):2376-2385. doi: 10.1016/j.ophtha.2016.07.032. Epub 2016 Sep 17. PMID 27651226
- [Background] Diabetic Retinopathy Clinical Research Network; Wells JA, Glassman AR, Ayala AR, Jampol LM, Aiello LP, Antoszyk AN, Arnold-Bush B, Baker CW, Bressler NM, Browning DJ, Elman MJ, Ferris FL, Friedman SM, Melia M, Pieramici DJ, Sun JK, Beck RW. Aflibercept, bevacizumab, or ranibizumab for diabetic macular edema. N Engl J Med. 2015 Mar 26;372(13):1193-203. doi: 10.1056/NEJMoa1414264. Epub 2015 Feb 18. PMID 25692915
- [Background] Wells JA, Glassman AR, Ayala AR, Jampol LM, Bressler NM, Bressler SB, Brucker AJ, Ferris FL, Hampton GR, Jhaveri C, Melia M, Beck RW; Diabetic Retinopathy Clinical Research Network. Aflibercept, Bevacizumab, or Ranibizumab for Diabetic Macular Edema: Two-Year Results from a Comparative Effectiveness Randomized Clinical Trial. Ophthalmology. 2016 Jun;123(6):1351-9. doi: 10.1016/j.ophtha.2016.02.022. Epub 2016 Feb 27. PMID 26935357
- [Background] Glassman AR, Wells JA 3rd, Josic K, Maguire MG, Antoszyk AN, Baker C, Beaulieu WT, Elman MJ, Jampol LM, Sun JK. Five-Year Outcomes after Initial Aflibercept, Bevacizumab, or Ranibizumab Treatment for Diabetic Macular Edema (Protocol T Extension Study). Ophthalmology. 2020 Sep;127(9):1201-1210. doi: 10.1016/j.ophtha.2020.03.021. Epub 2020 Mar 29. PMID 32402554
- [Background] Kim JE, Tomkins-Netzer O, Elman MJ, Lally DR, Goldstein M, Goldenberg D, Shulman S, Benyamini G, Loewenstein A. Evaluation of a self-imaging SD-OCT system designed for remote home monitoring. BMC Ophthalmol. 2022 Jun 10;22(1):261. doi: 10.1186/s12886-022-02458-z. PMID 35689210
- [Background] Liu Z, Huang W, Wang Z, Jin L, Congdon N, Zheng Y, Chen S, Liu Y. Evaluation of a self-imaging OCT for remote diagnosis and monitoring of retinal diseases. Br J Ophthalmol. 2024 Jul 23;108(8):1154-1160. doi: 10.1136/bjo-2023-324012. PMID 37903558
- [Background] Maguire MG, Liu D, Bressler SB, Friedman SM, Melia M, Stockdale CR, Glassman AR, Sun JK; DRCR Retina Network. Lapses in Care Among Patients Assigned to Ranibizumab for Proliferative Diabetic Retinopathy: A Post Hoc Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2021 Dec 1;139(12):1266-1273. doi: 10.1001/jamaophthalmol.2021.4103. PMID 34673898
- [Background] Greco G, Pistilli M, Asbell PA, Maguire MG; Dry Eye Assessment and Management Study Research Group. Association of Severity of Dry Eye Disease with Work Productivity and Activity Impairment in the Dry Eye Assessment and Management Study. Ophthalmology. 2021 Jun;128(6):850-856. doi: 10.1016/j.ophtha.2020.10.015. Epub 2020 Oct 15. PMID 33068617
- [Background] Bressler NM, Chang TS, Suner IJ, Fine JT, Dolan CM, Ward J, Ianchulev T; MARINA and ANCHOR Research Groups. Vision-related function after ranibizumab treatment by better- or worse-seeing eye: clinical trial results from MARINA and ANCHOR. Ophthalmology. 2010 Apr;117(4):747-56.e4. doi: 10.1016/j.ophtha.2009.09.002. Epub 2010 Mar 2. PMID 20189654
- [Result] Elman MJ, Ayala A, Bressler NM, Browning D, Flaxel CJ, Glassman AR, Jampol LM, Stone TW; Diabetic Retinopathy Clinical Research Network. Intravitreal Ranibizumab for diabetic macular edema with prompt versus deferred laser treatment: 5-year randomized trial results. Ophthalmology. 2015 Feb;122(2):375-81. doi: 10.1016/j.ophtha.2014.08.047. Epub 2014 Oct 28. PMID 25439614